CLINICAL TRIAL: NCT01661777
Title: Refractory Eustachian Tube Dysfunction: Are the Symptoms Related to Endolymphatic Hydrops?
Brief Title: Refractory Eustachian Tube Dysfunction: Are the Symptoms Related to Endolymphatic Hydrops
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Georges Wanna, assistant professor, Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JR08012012112856
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Eustachian Tube Dysfunction; Endolymphatic Hydrops
Keywords: Eustachian tube dysfunction; Endolymphatic hydrops; Diuretic; Low salt diet; Myringotomy; Pressure equalization tube; Ear tube; Ear fullness; Ear pressure; Allergy; Nasal steroid; Antihistamine
MeSH Terms: conditions — Endolymphatic Hydrops; Hypersensitivity | interventions — Diuretics; Histamine Antagonists; Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nasal steroid and Antihistamine (Other): Patients with ETD will be given nasal steroid and antihistamine for 8 weeks.
  Interventions: Drug: Nasal steroid; Drug: Antihistamine
- Myringotomy tubes (Active Comparator): Patients who fail nasal steroid and antihistamine treatment will have myringotomy tubes placed.
  Interventions: Procedure: Myringotomy tube placement
- Low salt diet and diuretic (Active Comparator): Patient's who fail to improve with myringotomy tubes will be treated with low salt det and diuretic
  Interventions: Drug: Diuretic; Behavioral: Low salt diet

INTERVENTIONS:
Drug: Nasal steroid
  Arms: Nasal steroid and Antihistamine
Procedure: Myringotomy tube placement
  Arms: Myringotomy tubes
Drug: Diuretic
  Arms: Low salt diet and diuretic
Drug: Antihistamine
  Arms: Nasal steroid and Antihistamine
Behavioral: Low salt diet
  Arms: Low salt diet and diuretic

SUMMARY:
The purpose of this study is to evaluate the benefit of treatment of refractory Eustachian tube dysfunction with standard treatment for endolymphatic hydrops. Eustachian tube dysfunction is a common diagnosis made in otolaryngology related to abnormal pressure equalization of the middle ear space related to a swollen, inflamed, or occluded Eustachian tube. The symptoms of this include perceived hearing loss, a feeling of fullness in the affected ear/ears, ear pain, ear popping, and occasionally imbalance. These symptoms overlap with a more rare and difficult to diagnose condition known as endolymphatic hydrops, or an overproduction to fluid in the inner ear. The treatment for these two conditions are distinct and traditionally, patients are treated for Eustachian tube dysfunction first as it is much more common and there are several treatments, namely nasal steroids, antihistamines, and pressure equalization tubes. For patients who do not improve with these treatments, they are often treated with diuretics and a low salt diet to treat for supposed endolymphatic hydrops. There has never been a study to investigate the utility of these treatments in patients with refractory Eustachian tube dysfunction. There is also reason to believe that chronic ETD with effusion can lead to both inner and middle ear dysfunction. Thus, this study aims to determine the benefit of standard endolymphatic hydrops treatment on patient with refractory Eustachian tube dysfunction symptoms in a prospective fashion.

Hypothesis:

Patients with refractory Eustachian tube dysfunction (patients with no or minimal symptom improvement despite nasal steroid and antihistamine treatment followed by myringotomy tube placement) have an element of endolymphatic hydrops and these patient's symptoms will improve with a low sodium diet and diuretic.

DETAILED DESCRIPTION:
Eustachian tube dysfunction is one of the most common problems encountered in general otolaryngology clinical practice. Symptoms of ear pressure, decreased hearing, ear pain, ear popping, and frequent ear infections are often blamed on the inability of the Eustachian tube to equalize air pressure across the ear drum. If the Eustachian tube is occluded, the middle ear space becomes a closed chamber in which normal gas exchange cannot occur. Treatment of Eustachian dysfunction has traditionally focused on a two tier system. First, patients are most often placed on a nasal steroid and an antihistamine. This medication regimen leads to decreased nasal inflammation, mucosal swelling, and treats nasal allergy. In many patients, this treatment improves symptoms completely or reduces them to a tolerable level. If the patient's symptoms are not improved, the next step in management is to create a surgical tract to the middle ear via a myringotomy (a hole across the ear drum) and placing a pressure equalization tube across the tympanic membrane. This bypasses any anatomical obstruction in the Eustachian tube and allows the middle ear pressure to equalize with the atmospheric pressure across the tympanic membrane. Unfortunately, despite this, there are patients with refractory symptoms, often ear pressure and subjectively decreased hearing. These symptoms are also frequently associated with inner ear disease, specifically endolymphatic hydrops. Endolymphatic hydrops is felt to be related to over production of endolymphatic fluid, the fluid within the inner ear. Thus, we propose that patient's will refractory Eustachian tube dysfunction are experiencing an inner ear phenomenon, and that they would benefit from treatment similar to how endolymphatic hydrops (or over production of endolymphatic fluid) is managed. The mainstays of management of endolymphatic hydrops are a low sodium diet and diuretic treatment (hydrochlorothiazide/triamterene). Both of these treatments aim to reduce endolymph production.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female patient 18-70 years old diagnosed with Eustachian tube dysfunction, as determined by clinical evaluation of symptoms and positive ETDQ-7.
* Non-smoker
* Normotensive or hypertensive (systolic blood pressure >115, diastolic blood pressure >75)
* Normal renal function (Cr <1.00)
* Not currently on acetazolamide
* Not currently on a low salt diet
* Competent in decision making process and able to sign a written informed consent form.
* No other previous alternative otologic diagnosis

Exclusion Criteria:

* Smoking
* Kidney disease (Cr >1.00)
* Hypotension (systolic blood pressure <115, diastolic blood pressure <75)
* Strong history of vascular disease (heart attack, stroke, heart failure, peripheral vascular disease i.e. claudication, gangrene, amputation)
* Alternative otologic diagnosis (Meniere's disease)
* Allergy or adverse reaction to previous administration of hydrochlorothiazide/triamterene
* Concurrent aspirin use
* Current or planned pregnancy during the course of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Improvement in patient ETD symptoms with nasal steroid and antihistamine alone | 2 years
  Determine the degree to which ETD symptoms are relieved with nasal steroid and antihistamine alone.
Improvement in patient ETD symptoms with pressure equalization tubes | 2 years
  Determine the degree to which patient's symptoms related to ETD improve after placement of pressure equalization tubes.
Improvement in patients with refractory ETD symptoms with treatment for endolymphatic hydrops with a diuretic and low salt diet | 2 years
  Determine the degree of improvement of patient symptoms in the setting of refractory ETD after a low salt diet and diuretic treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center--Division of Neurotology, Nashville, Tennessee, United States